CLINICAL TRIAL: NCT02851706
Title: Evaluation of the Natural History of and Specimen Banking for Patients With Tumors of the Central Nervous System
Brief Title: Natural History of and Specimen Banking for People With Tumors of the Central Nervous System
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160151; 16-C-0151
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-10-01

CONDITIONS: Brain Cancer; Brain Tumor; Spine Cancer; Spine Tumor; Neoplasm
Keywords: Brain Tumor; Glioma; Astrocytoma; Brain Cancer; Spine Cancer; Natural History
MeSH Terms: conditions — Brain Neoplasms; Spinal Cord Neoplasms; Neoplasms; Glioma; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First cohort Patients (Person with the disease): Patients with tumors of the central nervous system (CNS) who appear to be probable candidates for future protocol entry, have disease manifestations that are of unique scientific interest, importance, and/or educational value, or who have understudied tumors with unknown or unclear natural history. Patients with known genetic syndromes at high risk of developing CNS cancers will also be evaluated.
  Interventions: Other: No Treatment
- Second cohort Caregivers (Informants): Caregivers will be defined as anyone who patients identify as an unpaid close friend or family member who knows them well and who is involved with their day-to-day care.
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: No Treatment — Survey or Questionnaire Completion with or without Sample Submission

SUMMARY:
Background:

Brain and spinal cord tumors are uncommon. But they contribute substantially to cancer deaths in the U.S. in children and adults. Little progress has been made in treating brain tumors. Researchers want to learn more about these tumors by studying people who have them.

Objectives:

To understand brain and spinal cord tumors better and uncover areas for further research. Also, to connect people with these tumors to doctors who can help them manage their illness and give them new treatment options.

Design:

Participants will have an initial (baseline) visit. They will have their medical history taken and undergo physical and neurological exams. They will have blood tests. They may have scans (imaging studies) of the nervous system.

If participants have urine or cerebrospinal fluid collected during their regular care, researchers may save some.

Brain tumor tissue from a prior surgery may be studied.

Genomic DNA testing will be done on samples. Results will be linked to participants medical and/or family history.

The number of study visits at NIH will depend on the wishes of participants and their local doctors.

Participants will take a brain tumor survey on a computer. They can take it all at once or in 6 separate sections.

Participants will answer questions about their general well-being. They will answer questions to learn if they have symptoms of depression or anxiety.

Physicians will discuss test results with participants. They will recommend management and treatment options.

...

DETAILED DESCRIPTION:
Background:

This protocol is designed to meet an unmet need in neuro-oncology by evaluating patients with CNS tumors throughout their disease course. Data may be collected from multiple sources including medical records tests, and objective and subjective measures in patients and their caregivers. The protocol will evaluate patients with tumors of the central nervous system (CNS) who appear to be probable candidates for future protocol entry, have disease manifestations that are of unique scientific interest, importance, and/or educational value, or who have understudied tumors with unknown or unclear natural history. Patients with known genetic syndromes at high risk of developing CNS cancers will also be evaluated.

Objectives:

* To evaluate patients with tumors of the central nervous system (CNS) who are probable future candidates for NCI Phase I and II protocols.
* To follow patients with tumors of the CNS that are representative of important scientific and/or clinical principles
* To follow patients with CNS tumors that are understudied or have indeterminate natural history
* To evaluate and follow patients with known genetic syndromes at high risk of developing CNS cancers

Eligibility:

* All patients greater than or equal to 18 years of age with tumors of the CNS (or a history of tumors of the CNS) of interest to the NOB, who may be candidates for an NOB trial at some point in the future.
* Patients with tumors of the CNS that are of particular interest to members of the NOB because they pose important clinical and/or scientific questions and/or shed light on important aspects of the disease.
* Patients with known genetic syndromes at high risk of developing CNS cancers are eligible.
* Patients with rare tumors of the CNS who offer an important educational benefit to neuro-oncology trainees and staff.
* Caregivers, as identified by the patient are important to assess internal and external resources (e.g., coping mechanisms), identify specific factors that help patients with primary brain tumors face the uncertainty in their daily lives.
* Ability of patient or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

Design:

* All patients will undergo an initial evaluation by a member of the NOB or by a health care provider participating in the patient s care, where past medical and oncologic histories will be obtained as well as relevant data such as neuroimaging and pathology review. A total of 10,000 participants will be accrued to this study.
* Caregivers will be defined as anyone who patients identify as an unpaid close friend or family member who knows the NHS participant well and who is involved with their day-to-day care.
* Patients may be seen at the NIH Clinical Center at varying intervals depending on the clinical situation. Data related to the natural history of their disease course and outcome will be collected at least every visit at the NIH Clinical Center in which imaging is reviewed. Patients will be seen at a clinic visit or followed remotely at a minimum of once every year.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients (Person with the Disease)
* All patients >= 18 years of age with tumors of the CNS (or a history of tumors of the CNS) of interest to the NOB who may be future candidates for another NOB trial. This includes patients with undiagnosed imaging abnormalities in the central nervous system (brain and/or spinal cord) and patients with known genetic syndromes at high risk of developing CNS Cancers.
* Patients with tumors of the CNS that are of particular interest to members of the NOB because they pose important clinical and/or scientific questions and/or shed light on important aspects of the disease.
* Patients with rare tumors of the CNS (defined as occurring in less than 2,500 patients/year in the United States) who offer an important educational benefit to neuro-oncology trainees and staff.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
* Caregivers (Informants)
* Participants must be able to speak and read in English
* Age >= 18 years old
* Participant must be able to understand and willing to sign a written consent document
* Participants must be a caregiver for Natural History Study participants with the disease addressed above (Patients). Caregivers will be defined as anyone who patients identify as an unpaid close friend or family member who knows them well and who is involved with their day-to-day care.

EXCLUSION CRITERIA:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CNS Tumors and patients with known genetic syndromes at high risk of developing CNS cancers
Sampling Method: Non-Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
To evaluate patients with tumors of the central nervous system (CNS) who are probable future candidates for NCI Phase I and II protocols | completion of study
  Generalized knowledge about CNS tumors

CONTACTS AND LOCATIONS:
Overall Officials: Tito R Mendoza, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
BTRIS: All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@dbGaP: All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: BTRIS: Clinical data available during the study and indefinitely.@@@@@@dbGaP: Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: BTRIS: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@dbGaP: Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Stockdill ML, Vo JB, Celiku O, Kim Y, Karim Z, Vera E, Miller H, Gilbert MR, Armstrong TS. Neighborhood disadvantage is associated with treatment access outcomes and survival among individuals with a primary brain tumor. Neurooncol Pract. 2024 Nov 4;12(2):313-324. doi: 10.1093/nop/npae101. eCollection 2025 Apr. PMID 40110060
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0151.html